CLINICAL TRIAL: NCT02877797
Title: The Use of Cap Assisted Forward Viewing Esophagogastroduodenoscopy to Examine the Major Duodenal Papilla
Brief Title: Cap Assisted Upper Endoscopy to Visualize the Major Duodenal Papilla
Acronym: Kappa-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Monther Bajbouj, Prof. Dr. med., Technical University of Munich
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 14/16S
Record Dates: First submitted 2016-02-29; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Visualisation and Evaluation of Ampulla of Vater
MeSH Terms: interventions — Contraceptive Devices, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard Esophagogastroduodenoscopy (No Intervention): standard Esophagogastroduodenoscopy
- cap assisted Esophagogastroduodenoscopy (Experimental): cap assisted Esophagogastroduodenoscopy
  Interventions: Device: Cap

INTERVENTIONS:
Device: Cap — cap assisted esophagogastroduodenoscopy
  Arms: cap assisted Esophagogastroduodenoscopy

SUMMARY:
Aim of the present study is the evaluation of the diagnostic value of a cap assisted upper GI-endoscopy compared to a standard upper GI-endoscopy regarding the visualisation and evaluation of the papilla duodeni major.

ELIGIBILITY:
Inclusion Criteria:

* Indication of Esophagogastroduodenoscopy independent from the study
* Written informed
* Age ≥ 18 years

Exclusion Criteria:

* Absence of written informed consent
* Contraindication or absence of informed consent regarding sedation with Propofol
* Postoperativ changes of the upper GI-tract
* Intention of endoscopic intervention
* Suspicion of upper GI-bleeding
* Suspicion of stenosis of the esophagus
* Stent in the papilla duodeni major
* ASA (American Society of Anesthesiologists) classification ≥ 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Rate of complete visualisation of papilla duodeni major | 120 seconds
  visualisation: none, incomplete, complete

SECONDARY OUTCOMES:
Diagnostic yield in the upper GI-tract | up to 10 minutes
  All pathological findings which are seen during the examination should be reported (e.g. reflux esophagitis, Barret's esophagus, duodenal erosions, etc)
time of investigation | up to 10 minutes
  Duration of Esophagogastroduodenoscopy
complication rate | up to one week
  Any complications related to the examination within one week would be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan von Delius, Principal Investigator — Technical University of Munich
Locations (1):
- Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria, Germany